CLINICAL TRIAL: NCT04176679
Title: Diagnosis and Management of Enhanced Myometrial Vascularity Associated With Retained Products of Conception: a Retrospectif Moncentric Study
Brief Title: Diagnosis and Management of Enhanced Myometrial Vascularity Associated With Retained Products of Conception
Acronym: EMV RPOC AVM
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0532
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Hypervascularized Uterine Retentions
Keywords: Women; Retained Products of conception, Arterio venous malformation; color doppler ultrasound; embolization; fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Hypervascularized products of conception remain a topic debated in terms of definitions (ultrasound criteria, need complement by angio MRI) and management. The different uterine vascular lesions are often confused. This is a recurrent problem and care are heterogeneous. The aim of the study is to evaluate the management of these entities in CHU of Montpellier and determine more homogeneous care. The investigators further aimed to evaluate clinical presentation, ultrasound criteria, complications and the gynaecological and obstetrical outcomes of patients •Methods: This study will be conducted in compliance of ethic comitee. The investigators will collect data from 64 individuals, aged 18 to 50, suffering from uterine vascular lesions associated or not with products of conception between 2013 and 2019. Caracterisitics of the population, ultrasound and angio MRI data will be collected. Management wll be described as expectative, surgery or embolization of uterine arteries and the success or not will be noted. The investigators will question patients on their gynaecologic and obstetrical outcomes by telephone.

•Discussion: The investigators aim to define and characterize the different lesions, establish ultrasound criteria that would guide treatments. Describe the current treatments and compare them in terms of efficiency and safety in order to establish a homogeneous treatment protocol in our center

DETAILED DESCRIPTION:
* data are collected by computer software and patient phone calls
* ultrasounds criteria are reviewed by two clinicians
* statistical analysis is realized by a independent clinician
* the consent and agreement of the ethics committee has been sought

ELIGIBILITY:
Inclusion criteria:

* Women
* Aged between 18 and 50 years
* Managed in CHU Montpellier
* Diagnosis of hypervascularized products of conception
* Available ultrasound pictures

Exclusion criteria:

* Subject unable to understand the study
* Subject with another diagnosis of bleeding
* Subject who have retained products of conception with no vascularity or immediate curettage with uterine vacuity
* Subject who have no available ultrasound pictures

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women Aged between 18 and 50 years, and diagnosis of hypervascularized products of conception
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Evolution of the effects of the selected design products Evolution of the effects of the selected design products | 1 day
  the incidence of retained products of conception associated with enhanced myometrial vascularity
ultrasound vascularity assessment | 1 day
  ultrasound vascularity assessment for predicting future severe hemorrhage in retained products of conception with comparison of doppler color score (scale of the author Akiba, Kamaya and the Doppler color scoring system)
compare managing of these entities | 1 day
  compare managing of these entities: expectative, surgery, embolization, hysteroscopy in terms of efficiency (stopping bleeding) and safety

SECONDARY OUTCOMES:
assessment of the women quality of life | 1 day
  assessment of the women quality of life during managing , future fertility and pregnancy, gynaecologic healing with a telephone survey

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle VINTEJOUX, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC